CLINICAL TRIAL: NCT07041710
Title: Rehabilitation of Taste and Smell Disorders Associated With Chemotherapy Using Aromatherapy
Acronym: AGORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Médipôle Lyon-Villeurbanne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AGORA
Record Dates: First submitted 2025-06-04; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Taste

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): no taste and smell rehabilitation
  Interventions: Other: taste and smell disorders questionnaire
- experimental with day hospital (Experimental): During the day hospital, patients will be made aware of the various taste and smell disorders by the medical and paramedical team (doctor, dietician-nutritionist, speech therapist, therapeutic education nurse)
  Interventions: Other: experimental in day hospital; Other: taste and smell disorders questionnaire

INTERVENTIONS:
Other: experimental in day hospital — multidisciplinary day hospital
  Arms: experimental with day hospital
Other: taste and smell disorders questionnaire — Answer to the home-made questionnaire at inclusion and at 6 months

SUMMARY:
Changes in taste and smell can occur during chemotherapy treatment. These chemotherapy-related side effects can negatively impact patients' quality of life and diet.

The aim of this research is therefore to propose a solution to alleviate these taste and smell disorders. Based on the same principle as rehabilitation proposed for anosmia (loss of smell) related to COVID-19, we hypothesize that olfactory rehabilitation (using the sense of smell) through the odorous properties of essential oils could be effective for chemotherapy-related taste and smell alterations.

ELIGIBILITY:
Inclusion Criteria:

* cancer treated with chemotherapy
* patient with taste and/or smell disorders

Exclusion Criteria:

* patient at the end of chemotherapy treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
difference in scores between 6 months and the inclusion at "taste and smell disorders" questionnaire | 6 months
  taste and smell disorders home-made questionnaire (score from 0 to 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Médipôle Hôpital Mututaliste, Villeurbanne, France

IPD SHARING:
Plan to Share IPD: Undecided